CLINICAL TRIAL: NCT01666223
Title: Effect of Bile Acids in the Gut on GLP-1 Secretion in Healthy Subjects and Patients With Type 2 Diabetes
Brief Title: Effect of Bile Acids on GLP-1 Secretion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Morten Hansen, MD, PhD Student, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: H-1-2012-049
Record Dates: First submitted 2012-07-11; First posted 2012-08-16 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-12

CONDITIONS: Type 2 Diabetes; Obesity
Keywords: Type 2 diabetes; GLP-1; Bile acid; TGR-5
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Colesevelam Hydrochloride; Chenodeoxycholic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Colesevelam (Experimental)
  Interventions: Drug: Colesevelam
- Chenodeoxycholic acid (Experimental)
  Interventions: Drug: Chenodeoxycholic Acid
- Colesevelam + chenodeoxycholic acid (Experimental)
  Interventions: Drug: Colesevelam 3750 mg + chenodeoxycholic acid 1250 mg
- Placebo (Experimental)
  Interventions: Other: saline

INTERVENTIONS:
Drug: Colesevelam — Colesevelam 3750 mg dissolved in 100 ml saline, administered in a feeding tube at time = 0.
  Arms: Colesevelam
Drug: Chenodeoxycholic Acid — 1.250 mg dissolved in 100 ml saline, administered in a feeding tube at time = 0.
  Arms: Chenodeoxycholic acid
Other: saline — 100 ml saline
  Arms: Placebo
Drug: Colesevelam 3750 mg + chenodeoxycholic acid 1250 mg — Colesevelam and chenodeoxycholic acid dissolved in 100 ml saline, administered in a duodenal tube at time = 0.
  Arms: Colesevelam + chenodeoxycholic acid

SUMMARY:
The purpose of this study is to describe the physiological, pathophysiological and potentially therapeutic implications of bile-induced glucagon-like peptide-1 (GLP-1) secretion in human glucose homeostasis.

DETAILED DESCRIPTION:
The investigators hypothesize that even modest increments in endogenous GLP-1 secretion will elicit important antidiabetic effects of GLP-1. To evaluate whether bile acids have such effects, the investigators plan to perform intraduodenal infusion of two different bile acids and placebo.

ELIGIBILITY:
Patients with type 2 diabetes

Inclusion Criteria:

* danish caucasian ethnicity
* normal haemoglobin
* BMI > 25 kg/m2
* HbA1c < 9%
* informed consent

Exclusion Criteria:

* liver disease(ALT and AST > upper reference limit)
* gastrointestinal disease
* liver and biliary tract disease
* nephropathy (serum creatinine > 150 μM, and/or albuminuria)
* treatment with insulin, glp-1 analogues and/ or DPP-4 inhibitors
* treatment with medicine that can not be paused for 12 hours
* previous abdominal surgery eg. cholecystectomy
* BMI < 18,5 kg/m2 or > 35 kg/m2

Healthy Volunteers

Inclusion Criteria:

* danish caucasian ethnicity
* normal haemoglobin
* HbA1c < 6,0 (American Diabetes Association guidelines)
* informed consent

Exclusion Criteria:

* liver disease(ALT and AST > upper reference limit)
* gastrointestinal disease
* liver and biliary tract disease
* nephropathy (serum creatinine > 150 μM, and/or albuminuria)
* treatment with medicine that can not be paused for 12 hours
* previous abdominal surgery eg. cholecystectomy
* BMI < 18,5 kg/m2 or > 35 kg/m2
* first degree relatives diagnosed with diabetes
* previously diagnosed with diabetes, or treated with antidiabetic agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change in GLP-1 | At baseline, and at 5, 10, 20, 30, 40, 50, 60, 75, 90, 105, 120, 150 and 180 minutes

SECONDARY OUTCOMES:
Change in insulin | At baseline, and at 5, 10, 20, 30, 40, 50, 60, 75, 90, 105, 120, 150 and 180 minutes
Change in C-peptide | At baseline, and at 5, 10, 20, 30, 40, 50, 60, 75, 90, 105, 120, 150 and 180 minutes
Change in glucagon | At baseline, and at 5, 10, 20, 30, 40, 50, 60, 75, 90, 105, 120, 150 and 180 minutes
Change in glucagon-like-peptide 2 (GLP-2) | At baseline, and at 5, 10, 20, 30, 40, 50, 60, 75, 90, 105, 120, 150 and 180 minutes
Change in glucose-dependent insulinotropic polypeptide (GIP) | At baseline, and at 5, 10, 20, 30, 40, 50, 60, 75, 90, 105, 120, 150 and 180 minutes
Change in peptide YY (PYY) | At baseline, and at 5, 10, 20, 30, 40, 50, 60, 75, 90, 105, 120, 150 and 180 minutes
Change in oxyntomodulin | At baseline, and at 5, 10, 20, 30, 40, 50, 60, 75, 90, 105, 120, 150 and 180 minutes
Change in bile acids | At baseline, and at 5, 10, 20, 30, 40, 50, 60, 75, 90, 105, 120, 150 and 180 minutes
Change in gastrin | At baseline, and at 5, 10, 20, 30, 40, 50, 60, 75, 90, 105, 120, 150 and 180 minutes
Change in CCK | At baseline, and at 5, 10, 20, 30, 40, 50, 60, 75, 90, 105, 120, 150 and 180 minutes
Change in appetite, satiety and prospective food consumption | At baseline, and 30, 60, 90, 120 and 180 minutes
  Evaluated by Visual Analog Scale (VAS)
Change in gallbladder volume | -30, 0 (baseline), 30, 60, 120 og 180 minutes
  Evaluated by ultrasound
Change in basal metabolic rate | At -30, 60 og 150 minutes
  Evaluated by indirect calorimetry
Change in bile acid composition | At -30, 0, 30, 60, 120 og 180 minutes
  Evaluated by duodenal aspiration

CONTACTS AND LOCATIONS:
Overall Officials: Morten Hansen, MD, Principal Investigator — Diabetes Research Division, Department of Internal Medicine, Gentofte Hospital, University of Copenhagen
Locations (1):
- Diabetes Research Division, Department of Internal Medicine, Gentofte Hospital, University of Copenhagen, Hellerup, Copenhagen, Denmark

REFERENCES:
- [Background] Maruyama T, Miyamoto Y, Nakamura T, Tamai Y, Okada H, Sugiyama E, Nakamura T, Itadani H, Tanaka K. Identification of membrane-type receptor for bile acids (M-BAR). Biochem Biophys Res Commun. 2002 Nov 15;298(5):714-9. doi: 10.1016/s0006-291x(02)02550-0. PMID 12419312
- [Background] Adrian TE, Ballantyne GH, Longo WE, Bilchik AJ, Graham S, Basson MD, Tierney RP, Modlin IM. Deoxycholate is an important releaser of peptide YY and enteroglucagon from the human colon. Gut. 1993 Sep;34(9):1219-24. doi: 10.1136/gut.34.9.1219. PMID 8406158
- [Background] Katsuma S, Hirasawa A, Tsujimoto G. Bile acids promote glucagon-like peptide-1 secretion through TGR5 in a murine enteroendocrine cell line STC-1. Biochem Biophys Res Commun. 2005 Apr 1;329(1):386-90. doi: 10.1016/j.bbrc.2005.01.139. PMID 15721318
- [Background] Rafferty EP, Wylie AR, Hand KH, Elliott CE, Grieve DJ, Green BD. Investigating the effects of physiological bile acids on GLP-1 secretion and glucose tolerance in normal and GLP-1R(-/-) mice. Biol Chem. 2011 Apr;392(6):539-46. doi: 10.1515/BC.2011.050. Epub 2011 Apr 27. PMID 21521075